CLINICAL TRIAL: NCT05765162
Title: Safe Brain Initiative - Dedicated to Advancing Anaesthesia and Perioperative Personalised Care Towards Precision Anaesthesia Care. A Continuous Quality Improvement Initiative.
Brief Title: Safe Brain Initiative, Operationalizing Precision Anaesthesia
Acronym: SBI
Status: Recruiting | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Nykøbing Falster County Hospital (Other); Ankara University (Other); Naestved Hospital (Other); University of Bern (Other)
Responsible Party: Principal Investigator, Finn M. Radtke, Finn M. Radtke Ass. Professor, University of Southern Denmark
Other Study IDs: REG-117-2019
Record Dates: First submitted 2022-11-07; First posted 2023-03-13 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Neurocognitive Disorders; Post Operative Delirium; Pain; Nausea; Vomiting; Wellbeing; Shivering; Anxiety; Stress; Agitation,Psychomotor; Sedation Complication; Thirst; Satisfaction, Patient; Temperature Change, Body; Fasting; Sore-throat; Hearing and Vision Loss
MeSH Terms: conditions — Neurocognitive Disorders; Emergence Delirium; Pain; Nausea; Vomiting; Anxiety Disorders; Psychomotor Agitation; Patient Satisfaction; Body Temperature Changes; Fasting; Pharyngitis; Deaf-Blind Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients form age 18 and above: All patients form age 18 and above
  Interventions: Behavioral: Patient reported ourcomes

INTERVENTIONS:
Behavioral: Patient reported ourcomes — Full screening for the perioperative periode

SUMMARY:
Perioperatively, patients experience an unnecessarily high level of side effects associated with their treatment. These side effects include nausea, severe pain, anxiety, and stress. Moreover, many patients develop postoperative delirium (POD) and neurocognitive dysfunctions, often resulting in long-term cognitive impairment, decreased quality of life, and increased mortality. However, physicians, nurses and their institutions do not receive structured feedback regarding these aspects of each patient's well-being. They may therefore be unable to engage in the essential cause-and-effect learning necessary to evaluate and consecutively reduce such side effects.

Effective guidelines conform prevention is the proven key to shielding our patients from adverse Outcomes. The Safe Brain Initiative's high-quality routine data-for-action is a sword and accelerator for moving towards patient-centred, precision care. Thus, establishing a foundation for value-based and patient-centred healthcare development.

However, a turnkey real-world solution is challenging to develop and implement and requires substantial resources. As a result, such solutions are usually beyond the scope of a single institution. The SBI platform provides high-quality, real-world data to bridge this gap. It allows monitoring and in-depth analysis of cause and effect in the day-to-day routine of individuals, departments, and institutions.

The SBI's approach is continuously improved and updated. An organization called the SBI Global Society oversees the quality and precision of science through experts in the field. At SBI Hospitals and Flagship centres, Masterclasses are conducted and can be attended alongside clinical immersions.

SBI Solutions manages, develops, and provides technical and service support for the Safe Brain Initiative. Its service guarantees the professional and GDPR conform management of data handling and storage as well as the user-friendly functionality of the SBI-Dashboard solutions.

DETAILED DESCRIPTION:
The SBI core recommendations aim to monitor, detect and ultimately decrease and avoid the adverse side effects of surgery and anaesthesia in our daily routine care.Thereby guiding clinicians on the least invasive and least side effect-prone pathway through the perioperative process.Currently, the Safe Brain Initiative has 18 core recommendations available. All recommendations are non-invasive by nature, with the primary goal of detecting and preventing/reducing adverse outcomes.

SBI-Muda identifies both direct and derived economic effects. Despite being a central component of the broader SBI project, it also deserves and requires a specific focus. An inefficient OR management results in patient frustration, delays for the healthcare professionals, and a reduction in teamwork. Long waiting times can also increase stress and anxiety, prolong fluid fasting times, and exacerbate postoperative complications.

SBI-Muda will improve OR efficiency, reduce POD/PND, and improve patient-reported outcomes (PRO). By providing detailed SBI-Muda dashboard updates and feedback on OR and hospital metrics and placing them in context with the individual's outcomes (e.g., starting time or delay, suture to incision time, time spent in the postanaesthesia care unit (PACU) and postoperative time spent in the hospital). With SBI-Muda, the department as a whole and the healthcare specialist will have access to anonymized- more objective- systematized feedback on the quality of care and the metrics related to the perioperative process.

The SBI-Us functionality focuses on assessing the subjective quality of care provided by professional service providers (nurses, doctors, and other staff) and aligning this with patient-reported quality of care. In this regard, staff members will receive a brief anonymous questionnaire regarding their perception of treatment quality over the last three months. The results will be available to single health care professionals through SBI-me and the department as a whole.

SBI-Us provides a bidirectional perspective, including the patients' and the health care providers' perspectives, for benchmarking improvements in both areas and providing holistic, balanced information on the quality of care in the perioperative setting.

ELIGIBILITY:
Inclusion Criteria:

• All patients from age ≥18

Exclusion Criteria:

• All patients from age <18

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: • All surgical patients recieving anaesthesia from age ≥18
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | Perioperative
  Incidence of postoperative Delirium (Nu-DESC score 0-10) 0 is no delirium and 10 is highest delirium

SECONDARY OUTCOMES:
Patient reported outcome PRO´s | Perioperative
  Incidence of PONV (NRS 0-10) 10 is highest nausea 0 is no nausea / yes/no vomiting Incidence of Pain (NRS 0-10) 10 is highest pain 0 is no pain Incidence of Stress (NRS 0-10) 10 is highest stress 0 is no stress Incidence of Anxiety (NRS 0-10)) 10 is highest anxiety 0 is no anxiety Incidence of Sore throat (NRS 0-10) 10 is most sore 0 is no sore Incidents of Wellbeeing (NRS (0-10) 10 is best wellbeeing 0 is no wellbeeing Incidents of Shivering (NRS 0-10) 10 is highest shiviering 0 is no shivering Incidents of Thirst (NRS 0-10) 10 is highest thirst 0 is no thirst

CONTACTS AND LOCATIONS:
Overall Officials: Finn M. Radtke, Professor, Principal Investigator — University of Southern Denmark
Locations (1):
- Nykøbing Falster Hospital, Nykøbing Falster, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized patient outcome data (PRO´s)

REFERENCES:
- [Derived] Meco BC, Jakobsen K, De Robertis E, Buhre W, Alkis N, Kirkegaard PR, Hagi-Pedersen D, Bubser F, Koch S, Evered LA, Saunders SJ, Caterino M, Paolini F, Berger-Estilita J, Radtke FM. A first assessment of the safe brain initiative care bundle for addressing postoperative delirium in the postanesthesia care unit. J Clin Anesth. 2024 Oct;97:111506. doi: 10.1016/j.jclinane.2024.111506. Epub 2024 Jul 6. PMID 38972091